CLINICAL TRIAL: NCT00489970
Title: Persistence Study of GSK Biologicals' Tdap Vaccine (776423), 1, 3, 5 and 9 Years Following Administration as a Single Dose in NCT00346073 Study and to Evaluate the Immunogenicity and Safety of Boostrix as a Second Dose of Tdap, When Administered at Year 9
Brief Title: Persistence Study of GSK Biologicals' Tdap Vaccine 1, 3, 5 and 9 Years Following Administration as an Initial Single Dose in Healthy Young Adults and to Evaluate the Immunogenicity and Safety of Boostrix as a Second Dose of Tdap, When Administered at Year 9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110080; 110082 (Other: GSK); 110084 (Other: GSK); 110086 (Other: GSK)
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria
Keywords: Persistence; immunogenicity
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix; adacel

ARMS (3):
- Boostrix Group (Experimental): Subjects received in the primary study (NCT00346073) a single dose of Boostrix vaccine [Tdap](GSK776423) intramuscularly in the deltoid region of the non-dominant upper arm and in this study at Year 9 received a second dose of Boostrix vaccine [Tdap](GSK776423).
  Interventions: Procedure: Taking of blood samples; Biological: Boostrix
- Adacel Group (Active Comparator): Subjects received in the primary study (NCT00346073) a single dose of Adacel vaccine intramuscularly in the deltoid region of the non-dominant upper arm and in this study at Year 9 received a dose of Boostrix vaccine [Tdap](GSK776423).
  Interventions: Procedure: Taking of blood samples; Biological: Boostrix; Biological: Adacel
- Control group (Active Comparator): Subjects received the first dose of Boostrix vaccine [Tdap](GSK776423) in this study at Year 9.
  Interventions: Biological: Boostrix

INTERVENTIONS:
Procedure: Taking of blood samples — No treatment is planned to be given in this study. Blood samples will be collected at the following time points: 1 year, 3 years, 5 years and 9 years after the dose of vaccination.
  Arms: Adacel Group; Boostrix Group
Biological: Boostrix — A single dose of Boostrix was administered in the primary study (NCT00346073). No treatment was given in this study.
Biological: Adacel — A single dose of Adacel was administered in the primary study (NCT00346073). No treatment was given in this study.
  Arms: Adacel Group

SUMMARY:
The purpose of this study is to evaluate the persistence of antibodies against all the vaccine antigens 1, 3, 5 and 9 years after an initial vaccination with Tdap, and also to assess immunogenicity and safety of another dose of Boostrix, administered in this study.

This protocol posting deals with objectives and outcome measures of the extension phase. The objectives and outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00346073).

DETAILED DESCRIPTION:
Subjects were previously vaccinated with either Boostrix or a control Tdap vaccine (Sanofi Pasteurs' Adacel) in study NCT00346073. Only subjects who were part of the primary study will be invited to participate in this study. All subjects will receive a single dose of Boostrix at Visit 6 (Day 0) and subjects will be observed till Visit 7 (Day 30) for safety in terms of solicited adverse events (during 4 days post vaccination), unsolicited adverse events (during 31 days post vaccination) and serious adverse event (during the trial period). A blood sample will be collected from all subjects before vaccination (Visit 6) and one month after vaccination (Visit 7) for antibodies estimation.

This summary has been updated following Protocol amendment 1 dated 09 November 2010, amendment 2 dated 18 February 2014, and amendment 3 dated 10 December 2014. The protocol was amended first due to the following reasons:

1. The maximum window period allowed for the return of subjects for the Year 5 and Year 10 follow-up visits (Visit 5 and Visit 6) was extended from ± 5 weeks to ± 8 weeks.
2. The contact details for reporting of SAEs were clarified.
3. Text pertaining to the reporting of spontaneous abortion was removed from the protocol.
4. The number of attempts to contact subjects who did not return for scheduled persistence visits was clarified.

The main purpose of protocol amendment 2 is to evaluate the immunogenicity and safety of Boostrix as a second dose of Tdap vaccine when administered 8 years after an initial dose of Tdap. The Year 10 time point for evaluation of persistence has been cancelled because it is no longer feasible to conduct after a second dose of Tdap vaccine has been administered at Year 8.

The purpose of amendment 3 is to add co-primary objective to demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Boostrix group and Adacel group) is non-inferior to the immune response elicited by a first dose of Tdap vaccine (Control group), with respect to booster response against diphtheria, tetanus and pertussis (PT, FHA and PRN) antigens, one month following vaccination according to CBER's input. Accordingly, the study start has been pushed to Year 9 and this is reflected throughout the document.

ELIGIBILITY:
Inclusion Criteria:

• Persistence follow-up phase up to Year 9 time point:

The following criteria are applicable to subjects who refuse vaccination at Year 8 time point:

All subjects who received study vaccination (Boostrix or Adacel) in study NCT00346073 will be considered eligible to participate in this study.

Written informed consent must be obtained from the subject prior to each study time point.

Vaccination phase at Year 9 applicable for subjects in Boostrix and Adacel groups only:

The following criterion is applicable to subjects willing to consent to vaccination at Year 9 time point in the Boostrix and Adacel groups:

• All subjects who received study vaccination (Boostrix or Adacel) in study NCT00346073 will be considered eligible to participate in this study.

Vaccination phase at Year 9 applicable for subjects in the Control group only:

The following criterion is applicable to subjects willing to consent to vaccination at Year 9 time point in the Control group only:

• Subjects within the age range of 28-73 years will be considered eligible to participate in this study in the Control group.

Vaccination phase at Year 9 applicable for ALL subjects (Control, Boostrix and Adacel groups):

The following criteria are applicable to subjects willing to consent to vaccination at Year 9 time point in the Boostrix, Adacel and Control groups:

All subjects must satisfy the following criteria at study entry at Year 9 time point:

Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).

Written informed consent obtained from the subject for vaccination at Year 9 time point.

Healthy subjects as established by medical history and clinical examination before entering into the study.

* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of child bearing potential may be enrolled in the study, if the subject

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception for 1 month after completion of the vaccine dose

Exclusion Criteria:

The following criteria should be checked at the time of Year 9 vaccination time point. If any criteria is applicable, the subject must not be vaccinated in the study:

For subjects in Boostrix and Adacel groups:

• Administration of Tdap vaccine since the last dose received in the study NCT00346073.

For subjects in the Control group:

• Administration of Tdap (Boostrix or Adacel) vaccine at any time prior to the administration of Boostrix vaccine in this study.

For ALL subjects (Control, Boostrix and Adacel groups):

Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period, 31 days (Day 0-30).

* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to Visit 6 (pre-vacc). Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of vaccine, with the exception of inactivated Influenza vaccine which is allowed throughout the study period, 31 days (Day 0-30).

  -- Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Hypersensitivity to latex.
* History of diphtheria, tetanus or pertussis diseases.
* Severe allergic reaction (e.g. anaphylaxis) after previous administration of any tetanus toxoid, diphtheria toxoid, or pertussis-antigen containing vaccines, or any component of Boostrix.
* History of any neurological disorders or seizures.
* Encephalopathy (e.g. coma, decreased level of consciousness, prolonged seizures) of unknown etiology occurring within seven days following previous vaccination with pertussis-containing vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 100.4°F by any route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within three months preceding the dose of study vaccine or planned administration during the study period, 31 days (Day 0-30).

Administration of any tetanus or diphtheria containing vaccine or any registered or investigational vaccine utilizing a diphtheria toxoid or tetanus toxoid carrier within 5 years prior to the administration of Boostrix vaccine in this study.

* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions during the 31 day (Day 0-30) follow-up period post-vaccination.

Ages: 28 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1954 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2016-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (34):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, North Platte, Nebraska
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Grove City, Pennsylvania
  - GSK Investigational Site, Johnstown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=16064

REFERENCES:
- [Background] Brandon D, Kimmel M, Kuriyakose SO, Kostanyan L, Mesaros N. Antibody persistence and safety and immunogenicity of a second booster dose nine years after a first booster vaccination with a reduced antigen diphtheria-tetanus-acellular pertussis vaccine (Tdap) in adults. Vaccine. 2018 Oct 8;36(42):6325-6333. doi: 10.1016/j.vaccine.2018.08.051. Epub 2018 Sep 7. PMID 30197282
- [Derived] Weston W, Messier M, Friedland LR, Wu X, Howe B. Persistence of antibodies 3 years after booster vaccination of adults with combined acellular pertussis, diphtheria and tetanus toxoids vaccine. Vaccine. 2011 Nov 3;29(47):8483-6. doi: 10.1016/j.vaccine.2011.09.063. Epub 2011 Sep 25. PMID 21945698
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com
- See also: Redacted with child studies & included — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=110080&attachmentIdentifier=65724607-d004-4400-b36a-3fe9c67941ee&fileName=gsk-110080-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1592 participants were enrolled in the study at Year 1 (in the Boostrix and Adacel groups). As per advice from the Centre for Biologics and Research Evaluation (CBER), an additional treatment group acting as control was also added at Year 9, therefore the total number of subjects analyzed was 1592 (Year 1) + 362 (Year 9) = 1954.
Pre-assignment Details: Subjects who received a single dose of Boostrix or Adacel vaccines, in the primary study (NCT00346073) were included in this study.
Period: Persistence Year 1
Arm/Group | Boostrix Group | Adacel Group | Control Group
Started | 1069 | 523 | 0
Completed | 1069 | 523 | 0
Not Completed | 0 | 0 | 0
Period: Persistence Year 3
Arm/Group | Boostrix Group | Adacel Group | Control Group
Started | 1019 (Number of subjects who returned at Year 3) | 486 (Number of subjects who returned at Year 3) | 0
Completed | 1019 | 486 | 0
Not Completed | 0 | 0 | 0
Period: Persistence Year 5
Arm/Group | Boostrix Group | Adacel Group | Control Group
Started | 856 (Number of subjects who returned at Year 5) | 401 (Number of subjects who returned at Year 5) | 0
Completed | 856 | 401 | 0
Not Completed | 0 | 0 | 0
Period: Persistence Year 9
Arm/Group | Boostrix Group | Adacel Group | Control Group
Started | 309 (Number of subjects who returned at Year 9.) | 138 (Number of subjects who returned at Year 9.) | 362 (Number of subjects who received the first dose at Year 9.)
Completed | 306 | 136 | 357
Not Completed | 3 | 2 | 5
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Other | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Group | Adacel Group | Control Group | Total
Number analyzed (Participants) | 1069 | 523 | 362 | 1954
Age, Continuous [Mean (Standard Deviation); unit: years] — The data presented are the baseline values (Year 1 for Boostrix and Adacel groups and Year 9 for the Control Group).
  years | 41.7 (13.39) | 42.5 (13.27) | 52.0 (13.6) | 42.0 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants] — The data presented are the baseline values (Year 1 for Boostrix and Adacel groups and Year 9 for the Control Group).
  Participants
    Female | 680 | 357 | 196 | 1233
    Male | 389 | 166 | 166 | 721

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) Antibody Concentrations Greater Than or Equal to (≥) Protocol Specified Cut-off
Description: Anti-D cut-off was defined as ≥ 0.1 International Units per milliliter (IU/mL) determined with Enzyme-linked Immunosorbent Assay (ELISA)
Time Frame: At year 1 after the vaccination in primary study (NCT00346073)
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria and for whom data concerning immunogenicity endpoint measures obtained from the ATP cohort for immunogenicity corresponding to each time point were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1010 | 504
Participants | 967 | 489

2. Primary Outcome: Number of Subjects With Anti-D Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-D cut-off was defined as ≥ 0.1 IU/mL as assessed by ELISA
Time Frame: At year 3 after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 934 | 449
Participants | 857 | 425

3. Primary Outcome: Number of Subjects With Anti-D Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-D cut-off was defined as ≥ 0.1IU/mL as assessed by ELISA.
Time Frame: At year 5 after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 789 | 372
Participants | 735 | 359

4. Primary Outcome: Number of Subjects With Anti-D Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-D cut-off was defined as ≥ to 0.1IU/mL as assessed by ELISA.
Time Frame: At Year 9, one month before the booster vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 269 | 118
Participants | 245 | 113

5. Primary Outcome: Number of Subjects With Anti-tetanus (Anti-T) Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-T cut-off was defined as ≥ 0.1 IU/mL as assessed by ELISA.
Time Frame: At year 1 after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1014 | 506
Participants | 1000 | 504

6. Primary Outcome: Number of Subjects With Anti-T Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-T cut-off was defined as ≥ 0.1 IU/mL as assessed by ELISA.
Time Frame: At year 3 after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 937 | 442
Participants | 899 | 440

7. Primary Outcome: Number of Subjects With Anti-T Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-T cut-off was defined as ≥ 0.1 IU/mL as assessed by ELISA.
Time Frame: At year 5 after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 788 | 372
Participants | 772 | 370

8. Primary Outcome: Number of Subjects With Anti-T Antibody Concentrations ≥ Protocol Specified Cut-off
Description: Anti-T cut-off was defined as ≥ 0.1 IU/mL as assessed by ELISA.
Time Frame: At Year 9, one month before the booster vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 268 | 120
Participants | 263 | 120

9. Primary Outcome: Number of Subjects With Anti-D and Anti-T Concentrations ≥ 0.1 IU/mL and 1 IU/mL
Description: Number of subjects with anti-D and anti-T concentrations ≥ 0.1 IU/mL and 1 IU/mL were tabulated
Time Frame: At Year 9, one month after the booster vaccination.
Population: Analysis was performed on the According-to-Protocol (ATP) Cohort for analysis of immunogenicity at Year 9, which included all subjects who received the dose of study vaccine and for whom assay results were available for antibodies against at least one study vaccine antigen component after Year 9 vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 269 | 120 | 363
Participants
  Anti-D, ≥ 0.1 IU/ML: number analyzed (Participants) | 269 | 118 | 324
  Anti-D, ≥ 0.1 IU/ML | 245 | 113 | 265
  Anti-T, ≥ 0.1 IU/ML: number analyzed (Participants) | 268 | 120 | 324
  Anti-T, ≥ 0.1 IU/ML | 263 | 120 | 304
  Anti-D, ≥ 1 IU/ML: number analyzed (Participants) | 269 | 118 | 324
  Anti-D, ≥ 1 IU/ML | 114 | 54 | 92
  Anti-T, ≥ 1 IU/ML: number analyzed (Participants) | 268 | 120 | 324
  Anti-T, ≥ 1 IU/ML | 211 | 101 | 231
Statistical Analysis 1: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group and Control group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to seroprotection rate against diphtheria antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% confidence interval (CI) for the difference between groups in the seroprotection rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against diphtheria antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in percentage = 1.41, 97.5% CI 2-sided [-1.16 to 4.17] — Standardized asymptotic 97.5% CI for the group difference in the seroprotection rate was calculated
Statistical Analysis 2: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group and Control group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to seroprotection rate against tetanus antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% confidence interval (CI) for the difference between groups in the seroprotection rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against tetanus antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in percentage = 0.31, 97.5% CI 2-sided [-1.52 to 2.07] — Standardized asymptotic 97.5% CI for the group difference in the seroprotection rate was calculated
Statistical Analysis 3: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group and Control group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to seroprotection rate against diphtheria antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the seroprotection rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against diphtheria antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in percentage = 1.32, 97.5% CI 2-sided [-3.41 to 4.15] — Standardized asymptotic 97.5% CI for the group difference in the seroprotection rate was calculated
Statistical Analysis 4: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group and Control group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to seroprotection rate against tetanus antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the seroprotection rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against tetanus antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in percentage = 0.31, 97.5% CI 2-sided [-3.69 to 2.07] — Standardized asymptotic 97.5% CI for the group difference in the seroprotection rate was calculated

10. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations were measured by ELISA, tabulated as GMCs and expressed in IU/mL.
Time Frame: At Year 9, one month before booster vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 120 | 327
IU/mL
  Anti-PT | 8.2 [7.2 to 9.3] | 7.8 [6.5 to 9.4] | 5.4 [4.7 to 6.2]
  Anti-FHA | 42.2 [37.6 to 47.5] | 28.4 [24.0 to 33.4] | 23.6 [20.6 to 27.1]
  Anti-PRN: number analyzed (Participants) | 271 | 118 | 321
  Anti-PRN | 63.8 [53.1 to 76.7] | 64.7 [50.3 to 83.3] | 17.8 [14.7 to 21.6]

11. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations were measured by ELISA, tabulated as GMCs and expressed in IU/mL.
Time Frame: At Year 9, one month after the booster vaccination
Population: Analysis was performed on the Total Vaccinated Cohort (TVC) at Year 9 which included all subjects with a study vaccine administration dose documented: a safety analysis based on the TVC included all vaccinated subjects, an immunogenicity analysis based on the TVC included all vaccinated subjects for whom immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- Boostrix Group: Subjects received in the primary study (NCT00346073) a single dose of Boostrix vaccine [Tdap](GSK776423) intramuscularly in the deltoid region of the nondominant upper arm and in this study at Year 9 received a second dose of Boostrix vaccine [Tdap] (GSK776423).
- Adacel Group: Subjects received in the primary study (NCT00346073) a single dose of Adacel vaccine intramuscularly in the deltoid region of the non-dominant upper arm and in this study at Year 9 received a dose of Boostrix vaccine [Tdap](GSK776423) divided by Infanrix Group in APV-039 who included subjects who received 3 consecutive doses of Infanrix.
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 271 | 121
IU/mL
  ANTI-PT | 64.1 [56.8 to 72.3] | 70.4 [58.6 to 84.5]
  ANTI-FHA | 247.9 [227.3 to 270.3] | 254.6 [218.9 to 296.1]
  ANTI-PRN | 405.4 [359.3 to 457.5] | 511.8 [427.8 to 612.2]
Statistical Analysis 1: Comparison: Boostrix Group vs Adacel Group; To demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Boostrix Group) was non-inferior to the immune response elicited by a three dose series of Infanrix vaccine in infants in the German household contact efficacy study APV-039, with respect to antibodies against anti-PT one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limits of the 97.5% CIs for the anti-PT GMC ratios (Boostrix Group divided by Infanrix Group in APV-039) were greater than or equal to 0.67; GMC ratio; The associated CI was derived using the method proposed by G.Y. Zou and A. Donner [Zou, 2008]; GMC ratio = 1.53, 97.5% CI 2-sided [1.31 to 1.79]
Statistical Analysis 2: Comparison: Boostrix Group vs Adacel Group; To demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Boostrix Group) was non-inferior to the immune response elicited by a three dose series of Infanrix vaccine in infants in the German household contact efficacy study APV-039, with respect to antibodies against anti-FHA one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limits of the 97.5% CIs for the anti-FHA GMC ratios (Boostrix Group divided by Infanrix Group in APV-039) were greater than or equal to 0.67; GMC ratio; The associated CI was derived using the method proposed by G.Y. Zou and A. Donner [Zou, 2008]; GMC ratio = 5.27, 97.5% CI 2-sided [4.62 to 6.01]
Statistical Analysis 3: Comparison: Boostrix Group vs Adacel Group; To demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Boostrix Group) was non-inferior to the immune response elicited by a three dose series of Infanrix vaccine in infants in the German household contact efficacy study APV-039, with respect to antibodies against anti-PRN one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limits of the 97.5% CIs for the anti-PRN GMC ratios (Boostrix Group divided by Infanrix Group in APV-039) were greater than or equal to 0.67; GMC ratio; The associated CI was derived using the method proposed by G.Y. Zou and A. Donner [Zou, 2008]; GMC ratio = 3.62, 97.5% CI 2-sided [3.07 to 4.25]
Statistical Analysis 4: Comparison: Boostrix Group vs Adacel Group; To demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Adacel Group) was non-inferior to the immune response elicited by a three dose series of Infanrix vaccine in infants in the German household contact efficacy study APV-039, with respect to antibodies against anti-PT one month following vaccination; Test type: Non-Inferiority or Equivalence — One month after vaccination, the lower limits of the 97.5% CIs for the anti-PT GMC ratios (Adacel Group divided by Infanrix Group in APV-039) were greater than or equal to 0.67; GMC ratio; The associated CI was derived using the method proposed by G.Y. Zou and A. Donner [Zou, 2008]; GMC ratio = 1.64, 97.5% CI [1.33 to 2.03]
Statistical Analysis 5: Comparison: Boostrix Group vs Adacel Group; To demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Adacel Group) was non-inferior to the immune response elicited by a three dose series of Infanrix vaccine in infants in the German household contact efficacy study APV-039, with respect to antibodies against anti-FHA one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limits of the 97.5% CIs for the anti-FHA GMC ratios (Adacel Group divided by Infanrix Group in APV-039) were greater than or equal to 0.67; GMC ratio; The associated CI was derived using the method proposed by G.Y. Zou and A. Donner [Zou, 2008]; GMC ratio = 5.27, 97.5% CI 2-sided [4.37 to 6.36]
Statistical Analysis 6: Comparison: Boostrix Group vs Adacel Group; To demonstrate that the immune response elicited by a second dose of Tdap vaccine, Boostrix (Adacel Group) was non-inferior to the immune response elicited by a three dose series of Infanrix vaccine in infants in the German household contact efficacy study APV-039, with respect to antibodies against anti-PRN one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limits of the 97.5% CIs for the anti-PRN GMC ratios (Adacel Group divided by Infanrix Group in APV-039) were greater than or equal to 0.67; GMC ratio; The associated CI was derived using the method proposed by G.Y. Zou and A. Donner [Zou, 2008]; GMC ratio = 4.47, 97.5% CI 2-sided [3.58 to 5.57]

12. Primary Outcome: Booster Response to D and T Antigens
Description: A booster response was defined as: for initially seronegative subjects (S-) (pre-vaccination concentration below cut-off: < 0.1 IU/mL) antibody concentrations at least four times the cut-off (post vaccination concentration ≥ 0.4 IU/mL); for initially seropositive subjects (S+) (pre-vaccination concentration ≥ 0.1 IU/mL): an increase in antibody concentrations of at least four times the pre-vaccination concentration; Total = subjects either seropositive or seronegative.
Time Frame: At Year 9, one month after the booster vaccination.
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 269 | 120 | 324
Participants
  Anti-D, S-: number analyzed (Participants) | 24 | 5 | 58
  Anti-D, S- | 16 | 3 | 35
  Anti-D, S+: number analyzed (Participants) | 245 | 113 | 265
  Anti-D, S+ | 153 | 68 | 187
  Anti-D, Total: number analyzed (Participants) | 269 | 118 | 323
  Anti-D, Total | 169 | 71 | 222
  Anti-T, S-: number analyzed (Participants) | 5 | 0 | 20
  Anti-T, S- | 5 |  | 18
  Anti-T, S+: number analyzed (Participants) | 263 | 120 | 304
  Anti-T, S+ | 121 | 44 | 139
  Anti-T, Total: number analyzed (Participants) | 268 | 120 | 324
  Anti-T, Total | 126 | 44 | 157
Statistical Analysis 1: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against diphtheria antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against diphtheria antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -5.91, 97.5% CI 2-sided [-14.67 to 2.85] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 2: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against tetanus antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against tetanus antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -1.44, 97.5% CI 2-sided [-10.63 to 7.79] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 3: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against diphtheria antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against diphtheria antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -8.56, 97.5% CI 2-sided [-20.33 to 2.73] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 4: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against tetanus antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against tetanus antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -11.79, 97.5% CI 2-sided [-22.98 to 0.15] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated

13. Primary Outcome: Booster Response to PT, FHA and PRN Antigens
Description: Booster response was defined as: for subjects with pre-vaccination antibody concentration < 5 EL.U/mL (S-): antibody concentration ≥ 20 EL.U/mL; for subjects with pre-vaccination antibody concentration ≥ 5 EL.U/mL and < 20 EL.U/mL (S+, <4*cut-off): antibody concentration at least four times the pre-vaccination concentration; for subjects with pre-vaccination antibody concentration ≥ 20 EL.U/mL (S+, ≥4*cut-off): antibody concentration at least two times the pre-vaccination concentration; Total = subjects either seropositive or seronegative
Time Frame: At Year 9, one month after the booster vaccination.
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 120 | 327
Participants
  Anti-PT, S-: number analyzed (Participants) | 41 | 14 | 117
  Anti-PT, S- | 34 | 10 | 101
  Anti-PT, S+, < 4*cut-off: number analyzed (Participants) | 124 | 60 | 104
  Anti-PT, S+, < 4*cut-off | 106 | 53 | 94
  Anti-PT, S+, ≥ 4*cut-off: number analyzed (Participants) | 106 | 46 | 105
  Anti-PT, S+, ≥ 4*cut-off | 95 | 43 | 97
  Anti-PT, Total: number analyzed (Participants) | 271 | 120 | 326
  Anti-PT, Total | 235 | 106 | 292
  Anti-FHA, S-: number analyzed (Participants) | 0 | 1 | 5
  Anti-FHA, S- |  | 1 | 5
  Anti-FHA, S+, < 4*cut-off: number analyzed (Participants) | 16 | 9 | 71
  Anti-FHA, S+, < 4*cut-off | 16 | 9 | 70
  Anti-FHA, S+, ≥ 4*cut-off: number analyzed (Participants) | 255 | 110 | 251
  Anti-FHA, S+, ≥ 4*cut-off | 216 | 106 | 228
  Anti-FHA, Total | 232 | 116 | 303
  Anti-PRN, S-: number analyzed (Participants) | 4 | 1 | 37
  Anti-PRN, S- | 4 | 1 | 31
  Anti-PRN, S+, < 4*cut-off: number analyzed (Participants) | 29 | 10 | 78
  Anti-PRN, S+, < 4*cut-off | 27 | 10 | 75
  Anti-PRN, S+, ≥ 4*cut-off: number analyzed (Participants) | 238 | 107 | 205
  Anti-PRN, S+, ≥ 4*cut-off | 179 | 87 | 175
  Anti-PRN, Total: number analyzed (Participants) | 271 | 118 | 320
  Anti-PRN, Total | 210 | 98 | 281
Statistical Analysis 1: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against PT antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against PT antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -2.85, 97.5% CI 2-sided [-9.09 to 3.08] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 2: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against FHA antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against FHA antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -7.05, 97.5% CI 2-sided [-13.16 to -1.40] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 3: Comparison: Boostrix Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Boostrix group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against PRN antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Boostrix group) minus the first dose of Boostrix (Control group)] against PRN antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -10.32, 97.5% CI 2-sided [-17.50 to -3.38] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 4: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against PT antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against PT antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = -1.24, 97.5% CI 2-sided [-10.03 to 5.57] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 5: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against FHA antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against FHA antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response rate = 4.01, 97.5% CI 2-sided [-2.38 to 8.66] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated
Statistical Analysis 6: Comparison: Adacel Group vs Control Group; To demonstrate that the immune response elicited by a second dose of Boostrix vaccine (Adacel group) was non-inferior to the immune response elicited by a first dose of Boostrix vaccine (Control group), with respect to booster response against PRN antigen, one month following vaccination; Test type: Non-Inferiority — One month after vaccination, the lower limit of the 97.5% CI for the difference between groups in the booster response rate [a second dose of Boostrix (Adacel group) minus the first dose of Boostrix (Control group)] against PRN antigen was greater than or equal to -10% (clinical limit for non-inferiority); Difference in booster response = -4.76, 97.5% CI 2-sided [-14.53 to 3.18] — Standardized asymptotic 97.5% CI for the group difference in the Booster response was calculated

14. Secondary Outcome: Number of Subjects With Anti-pertussis Toxoid (PT) Antibody Concentrations Equal to or Above Protocol Specified Cut-off
Description: The cut-off for anti-PT concentrations was defined as ≥ 5 ELISA units per mililiter (EL.U/mL).
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1013 | 506
Participants
  Year 1 | 917 | 435
  Year 3: number analyzed (Participants) | 914 | 442
  Year 3 | 751 | 316
  Year 5: number analyzed (Participants) | 790 | 372
  Year 5 | 670 | 285

15. Secondary Outcome: Number of Subjects With Anti-PT Antibody Concentrations Equal to or Above Protocol Specified Cut-off
Description: The cut-off for anti-PT concentrations was defined as equal to or greater than 2.693 IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 327
Participants
  Pre-booster: number analyzed (Participants) | 271 | 120 | 327
  Pre-booster | 230 | 106 | 209
  Post-booster: number analyzed (Participants) | 271 | 121 | 326
  Post-booster | 268 | 120 | 322

16. Secondary Outcome: Number of Subjects With Anti-FHA Antibody Concentrations Equal to or Above Protocol Specified Cut-off
Description: The cut-off for anti-FHA concentrations was defined as equal to or greater than 5 EL.U/mL.
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1014 | 502
Participants
  Year 1 | 1012 | 501
  Year 3: number analyzed (Participants) | 916 | 439
  Year 3 | 913 | 437
  Year 5: number analyzed (Participants) | 789 | 371
  Year 5 | 788 | 368

17. Secondary Outcome: Number of Subjects With Anti-FHA Antibody Concentrations Equal to or Above Protocol Specified Cut-off
Description: The cut-off for anti-FHA concentrations was defined as equal to or greater than 2.046 IU/mL
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 327
Participants
  Pre-booster: number analyzed (Participants) | 271 | 120 | 327
  Pre-booster | 271 | 119 | 322
  Post-booster | 271 | 121 | 327

18. Secondary Outcome: Number of Subjects With Anti-PRN Antibody Concentrations Equal to or Above Protocol Specified Cut-off
Description: The cut-off for anti-PRN concentrations was defined as equal to or greater than 5 EL.U/mL.
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1011 | 501
Participants
  Year 1 | 971 | 489
  Year 3: number analyzed (Participants) | 915 | 442
  Year 3 | 862 | 426
  Year 5: number analyzed (Participants) | 782 | 371
  Year 5 | 755 | 362

19. Secondary Outcome: Number of Subjects With Anti-PRN Antibody Concentrations Equal to or Above Protocol Specified Cut-off
Description: The cut-off for anti-PRN concentrations was defined as equal to or greater than 2.187 IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 326
Participants
  Pre-booster: number analyzed (Participants) | 271 | 118 | 321
  Pre-booster | 267 | 117 | 284
  Post-booster | 271 | 121 | 326

20. Secondary Outcome: Anti-D Antibody Concentration
Description: Anti-D antibody concentration is expressed as geometric mean concentration (GMC) in IU/mL.
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1010 | 504
IU/mL
  Year 1 | 1.4 [1.3 to 1.6] | 1.4 [1.3 to 1.6]
  Year 3: number analyzed (Participants) | 914 | 442
  Year 3 | 0.9 [0.8 to 1.0] | 1.0 [0.9 to 1.1]
  Year 5: number analyzed (Participants) | 789 | 372
  Year 5 | 0.8 [0.7 to 0.9] | 0.9 [0.8 to 1.0]

21. Secondary Outcome: Anti-D Antibody Concentration
Description: Anti-D antibody concentration is expressed as GMC in IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 326
IU/mL
  Pre-booster: number analyzed (Participants) | 269 | 118 | 324
  Pre-booster | 0.7 [0.6 to 0.8] | 0.8 [0.6 to 0.9] | 0.4 [0.4 to 0.5]
  Post-booster | 4.1 [3.6 to 4.7] | 4.7 [3.9 to 5.7] | 4.0 [3.4 to 4.6]

22. Secondary Outcome: Anti-T Antibody Concentration
Description: Anti-T antibody concentration is expressed as GMC in IU/mL.
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1014 | 506
IU/mL
  Year 1 | 3.4 [3.2 to 3.6] | 4.4 [4.1 to 4.7]
  Year 3: number analyzed (Participants) | 917 | 442
  Year 3 | 2.2 [2.1 to 2.3] | 2.9 [2.7 to 3.1]
  Year 5: number analyzed (Participants) | 788 | 372
  Year 5 | 2.0 [1.9 to 2.1] | 2.5 [2.3 to 2.7]

23. Secondary Outcome: Anti-T Antibody Concentration
Description: Anti-T antibody concentration is expressed as GMC in IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 327
IU/mL
  Pre-booster: number analyzed (Participants) | 268 | 120 | 324
  Pre-booster | 1.8 [1.6 to 2.0] | 2.3 [2.0 to 2.7] | 1.5 [1.3 to 1.7]
  Post-booster | 8.4 [7.7 to 9.3] | 8.6 [7.6 to 9.8] | 8.8 [8.0 to 9.7]

24. Secondary Outcome: Anti-PT Antibody Concentration
Description: Anti-PT antibody concentration is expressed as GMC in EL.U/mL.
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1013 | 506
IU/mL
  Year 1 | 22.4 [21.0 to 24.0] | 15.6 [14.2 to 17.2]
  Year 3: number analyzed (Participants) | 914 | 442
  Year 3 | 14.1 [13.0 to 15.0] | 10.0 [9.0 to 11.1]
  Year 5: number analyzed (Participants) | 790 | 372
  Year 5 | 14.6 [13.5 to 15.8] | 11.6 [10.3 to 13.0]

25. Secondary Outcome: Anti-PT Antibody Concentration
Description: Anti-PT antibody concentration was expressed as GMC in IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 327
IU/mL
  Pre-booster: number analyzed (Participants) | 271 | 120 | 327
  Pre-booster | 8.2 [7.2 to 9.3] | 7.8 [6.5 to 9.4] | 5.4 [4.7 to 6.2]
  Post-booster: number analyzed (Participants) | 271 | 121 | 326
  Post-booster | 64.1 [56.8 to 72.3] | 70.4 [58.6 to 84.5] | 66.2 [58.5 to 74.8]

26. Secondary Outcome: Anti-FHA Antibody Concentration
Description: Anti-FHA antibody concentration is expressed as GMC in IU/mL
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1014 | 502
IU/mL
  Year 1 | 190.1 [178.5 to 202.6] | 118.8 [108.7 to 129.9]
  Year 3: number analyzed (Participants) | 916 | 439
  Year 3 | 114.1 [107.1 to 121.5] | 81.8 [74.7 to 89.4]
  Year 5: number analyzed (Participants) | 789 | 371
  Year 5 | 110.0 [103.0 to 117.4] | 80.8 [73.1 to 89.4]

27. Secondary Outcome: Anti-FHA Antibody Concentration
Description: Anti-FHA antibody concentration was expressed as GMC in IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 327
IU/mL
  Pre-booster: number analyzed (Participants) | 271 | 120 | 327
  Pre-booster | 42.2 [37.6 to 47.5] | 28.4 [24.0 to 33.4] | 23.6 [20.6 to 27.1]
  Post-booster | 247.9 [227.3 to 270.3] | 254.6 [218.9 to 296.1] | 373.6 [336.5 to 414.8]

28. Secondary Outcome: Anti-PRN Antibody Concentration
Description: Anti-PRN antibody concentration is expressed as GMC in IU/mL
Time Frame: At 1, 3, and 5 years after the vaccination in primary study (NCT00346073)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group
Number analyzed (Participants) | 1011 | 501
IU/mL
  Year 1 | 152.2 [137.2 to 168.8] | 132.5 [115.6 to 151.8]
  Year 3: number analyzed (Participants) | 915 | 442
  Year 3 | 82.5 [74.4 to 91.5] | 70.6 [61.6 to 81.0]
  Year 5: number analyzed (Participants) | 782 | 371
  Year 5 | 85.3 [76.7 to 94.9] | 77.4 [66.9 to 89.6]

29. Secondary Outcome: Anti-PRN Antibody Concentration
Description: Anti-PRN antibody concentration is expressed as GMC in IU/mL.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 326
IU/mL
  Pre-booster: number analyzed (Participants) | 271 | 118 | 321
  Pre-booster | 63.8 [53.1 to 76.7] | 64.7 [50.3 to 83.3] | 17.8 [14.7 to 21.6]
  Post-booster | 405.4 [359.3 to 457.5] | 511.8 [427.8 to 612.2] | 336.4 [283.3 to 399.4]

30. Secondary Outcome: Alternative Booster Response to Anti-D and Anti-T Antigens
Description: Alternative Booster response to D and T antigens is defined as: - For subjects with pre-booster antibody concentration below 0.1 IU/mL: antibody concentrations at least four times the 0.1IU/ML, one month after vaccination, and - For subjects with pre-booster antibody concentration ≥0.1 IU/mL and <1.0 IU/mL: antibody concentrations of at least four times the pre-booster antibody concentration, one month after vaccination. - For subjects with pre-booster antibody concentration ≥1.0 IU/mL and <6.0 IU/mL: antibody concentrations of at least two times the pre-booster antibody concentration, one month after vaccination. - Subjects with pre-booster antibody concentration ≥6.0 IU/mL are not evaluable for booster response. S- = Antibody concentration < 0.1 IU/mL S+ = Antibody concentration ≥ 0.1 IU/mL Total = subjects either seropositive or seronegative
Time Frame: At Year 9, one month after booster vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 259 | 115 | 311
Participants
  ANTI-D, S-: number analyzed (Participants) | 24 | 5 | 58
  ANTI-D, S- | 16 | 3 | 35
  ANTI-D, S+ (<1 IU/ML): number analyzed (Participants) | 131 | 59 | 173
  ANTI-D, S+ (<1 IU/ML) | 103 | 45 | 148
  ANTI-D, S+ (≥1 IU/ML): number analyzed (Participants) | 104 | 51 | 80
  ANTI-D, S+ (≥1 IU/ML) | 84 | 40 | 65
  ANTI-D, Total | 203 | 88 | 248
  ANTI-T, S-: number analyzed (Participants) | 5 | 0 | 20
  ANTI-T, S- | 5 |  | 18
  ANTI-T, S+ (<1 IU/ML): number analyzed (Participants) | 52 | 19 | 73
  ANTI-T, S+ (<1 IU/ML) | 46 | 14 | 65
  ANTI-T, S+ (≥1 IU/ML): number analyzed (Participants) | 191 | 92 | 196
  ANTI-T, S+ (≥1 IU/ML) | 151 | 74 | 159
  ANTI-T, Total: number analyzed (Participants) | 248 | 111 | 289
  ANTI-T, Total | 202 | 88 | 242

31. Secondary Outcome: Alternative Booster Responses to Anti-PT, Anti-FHA and Anti-PRN Antigens
Description: Alternative Booster response to PT, FHA and PRN antigens is defined as: - For subjects with pre-booster antibody concentration below the assay cut off: antibody concentrations at least four times the assay cut off one month after vaccination, and - For subjects with pre-booster antibody concentration ≥ assay cut off and < 60 IU/mL: antibody concentration increase of at least 30 IU/mL from the pre-booster antibody concentration, one month after vaccination. - For subjects with pre-booster antibody concentration ≥ 60 IU/mL : at least 1.5 fold increase of antibody concentration from the pre-booster antibody concentration, one month after vaccination. S- = seronegative subjects (antibody concentration below assay cut off for anti-PT, anti-FHA, anti-PRN) S+ = seropositive subjects (antibody concentration below assay cut off for anti-PT, anti-FHA, anti-PRN) Total = subjects either seropositive or seronegative
Time Frame: At Year 9, one month after booster vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 120 | 327
Participants
  ANTI-FHA, S-: number analyzed (Participants) | 0 | 1 | 5
  ANTI-FHA, S- |  | 1 | 5
  ANTI-FHA, ≥ assay Cut-off and < 60 IU/mL: number analyzed (Participants) | 174 | 91 | 245
  ANTI-FHA, ≥ assay Cut-off and < 60 IU/mL | 171 | 91 | 241
  ANTI-FHA, ≥ 60 IU/mL: number analyzed (Participants) | 97 | 28 | 77
  ANTI-FHA, ≥ 60 IU/mL | 82 | 27 | 64
  ANTI-FHA, Total | 253 | 119 | 310
  ANTI-PRN, S-: number analyzed (Participants) | 4 | 1 | 37
  ANTI-PRN, S- | 4 | 1 | 31
  ANTI-PRN, ≥ assay Cut-off and < 60 IU/mL: number analyzed (Participants) | 118 | 53 | 200
  ANTI-PRN, ≥ assay Cut-off and < 60 IU/mL | 115 | 52 | 185
  ANTI-PRN, ≥ 60 IU/mL: number analyzed (Participants) | 149 | 64 | 83
  ANTI-PRN, ≥ 60 IU/mL | 111 | 53 | 62
  ANTI-PRN, Total: number analyzed (Participants) | 271 | 118 | 320
  ANTI-PRN, Total | 230 | 106 | 278
  ANTI-PT, S-: number analyzed (Participants) | 41 | 14 | 117
  ANTI-PT, S- | 34 | 10 | 101
  ANTI-PT, ≥ assay Cut-off and < 60 IU/mL: number analyzed (Participants) | 222 | 103 | 194
  ANTI-PT, ≥ assay Cut-off and < 60 IU/mL | 169 | 83 | 166
  ANTI-PT, ≥ 60 IU/mL: number analyzed (Participants) | 8 | 3 | 15
  ANTI-PT, ≥ 60 IU/mL | 7 | 3 | 10
  ANTI-PT, Total: number analyzed (Participants) | 271 | 120 | 326
  ANTI-PT, Total | 210 | 96 | 277

32. Secondary Outcome: Seroprotection Status for Anti-D Antibody Concentration
Description: Seroprotection status for anti-D antibody concentration < 0.1 IU/mL were tested for neutralizing antibodies using a VERO-cell neutralization assay. Seroprotection rate is defined as the percentage of subjects with antibody concentrations greater than or equal (≥) the seroprotection cut-off value defined for that antibody.
Time Frame: At Year 9, one month before(pre booster) and after the booster vaccination(post booster)
Population: as for outcome 9
Measure: Number; unit: Percentage of subjects
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 271 | 121 | 326
Percentage of subjects
  Pre-booster: number analyzed (Participants) | 269 | 118 | 324
  Pre-booster | 8.3 | 40.0 | 27.6
  Post-booster | 50.0 | 0.0 | 14.3

33. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Year 9
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as significant pain at rest that prevented normal everyday activities. Grade 3 redness and swelling was greater than 50 millimeters (mm)
Time Frame: During the 4-day (Days 0-3) post vaccination period.
Population: The analysis was performed on the Total Vaccinated cohort at Year 9, which included all subjects with study vaccine administration dose documented, who returned at Year 9 and had their diary cards completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 306 | 137 | 358
Participants
  Any Pain | 180 | 84 | 132
  Grade 3 Pain | 3 | 1 | 4
  Any Redness | 74 | 32 | 53
  Grade 3 Redness | 5 | 2 | 0
  Any Swelling | 57 | 26 | 41
  Grade 3 Swelling | 4 | 2 | 2

34. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms - Year 9
Description: The solicited general symptoms assessed were Fatigue, Gastrointestinal symptoms (including nausea, vomiting, diarrhea and abdominal pain), Headache and Fever [defined as temperature of ≥100.4 degrees Fahrenheit (F) by any route]. Any = Occurrence of any general symptom regardless of its intensity grade or relationship to vaccination; Grade 3 Symptom = Symptom that prevented normal activity; Grade 3 Fever > 104.0 degrees F.
Time Frame: During the 4-day (Days 0-3) post vaccination period.
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 306 | 137 | 358
Participants
  Any Fatigue | 71 | 23 | 51
  Grade 3 Fatigue | 3 | 1 | 0
  Any Gastrointestinal symptoms | 27 | 4 | 29
  Grade 3 Gastrointestinal symptoms | 0 | 0 | 0
  Any Headache | 52 | 25 | 53
  Grade 3 Headache | 0 | 1 | 1
  Any Fever | 2 | 0 | 2
  Grade 3 Fever | 0 | 0 | 0

35. Secondary Outcome: Number of Subjects With Any Large Injection Site Reaction - Year 9
Description: Large injection site reaction = a swelling with a diameter > 100 mm, noticeable diffuse swelling or noticeable increase in limb circumference.
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort at Year 9, which included all subjects with study vaccine administration dose documented, who returned at Year 9.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 309 | 138 | 362
Participants | 0 | 0 | 0

36. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - Year 9
Description: An unsolicited AE covers any untoward medical oc-currence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Days 0-30) post-vaccination period.
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Groups:
- Adacel Group: Subjects received in the primary study (NCT00346073) a single dose of Adacel vaccine intramuscularly in the deltoid region of the non-dominant upper arm.
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 309 | 138 | 362
Participants | 42 | 23 | 37

37. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - Year 9
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group | Adacel Group | Control Group
Number analyzed (Participants) | 309 | 138 | 362
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day post-vaccination period; Unsolicited AE(s): during the 31-day (Day 0-30) post vaccination period; SAE(s): during the 31-day (Day 0-30) post vaccination period
Description: Safety data is presented for subjects who received the study vaccine (at year 9) in this study.
Arm/Group | Boostrix Group | Adacel Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/309 | 0/138 | 0/362
Serious Adverse Events (participants affected / at risk) | 0/309 | 0/138 | 1/362
Other Adverse Events (participants affected / at risk) | 213/309 | 95/138 | 172/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Group (N=309) | Adacel Group (N=138) | Control Group (N=362)
Seizure (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Group (N=309) | Adacel Group (N=138) | Control Group (N=362)
Gastrointestinal disorder (Gastrointestinal disorders) | 28 (28) | 4 (4) | 29 (29)
Fatigue (General disorders) | 71 (72) | 23 (23) | 51 (51)
Pain (General disorders) | 181 (183) | 84 (84) | 132 (132)
Swelling (General disorders) | 57 (57) | 26 (26) | 41 (41)
Headache (Nervous system disorders) | 53 (54) | 28 (29) | 57 (58)
Erythema (Skin and subcutaneous tissue disorders) | 74 (74) | 32 (32) | 53 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.